CLINICAL TRIAL: NCT00289263
Title: Maintenance Paclitaxel Vs Control After Anthracycline/Paclitaxel Combined First-Line Chemotherapy in Metastatic Breast Cancer
Brief Title: Maintenance Chemotherapy in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MANTA 1 Study Italian Collaborative Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANTA1
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2003-11

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; maintenance chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel

SUMMARY:
This is a randomized, prospective and multicenter phase III study. Two-hundred-sixty-two (262) patients on each arm will be recruited in the study.

DETAILED DESCRIPTION:
The primary objective is time to disease progression. All patients must be treated with first line chemotherapy, consisting of one of the following regimens: a) ET (epirubicin 90 mg/sqm day 1 plus paclitaxel 200 mg/sqm (3 hour infusion) day 1, or b) AT (doxorubicin 50 mg/sqm day 1 plus paclitaxel 200 mg/sqm (3 hour infusion) day 2, administered on a 3 weekly schedule.

Patients with complete response, partial response or stable disease are eligible for MANTA1 study.

The expected median progression free survival of metastatic breast cancer patients who achieve a disease control after first line chemotherapy was estimated to be 10 months. The minimal improvement, justifying the adoption of maintenance paclitaxel, was estimated to be at least 3 months. With 262 eligible patients on each arm, the trial will have a power of 80% to detect a 30% improvement in median progression free survival, testing at the two-sided .05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients with metastatic breast cancer in response or stable disease after six to eight courses of first line induction chemotherapy treatment
* Measurable and/or evaluable disease
* Performance status ECOG 0, 1, 2.
* Normal cardiac function, confirmed by left ventricular ejection fraction (LVEF).

Exclusion Criteria:

* Presence of peripheral neuropathy > grade 2 by NCI Common Toxicity Criteria (NCI-CTC) following induction chemotherapy
* Adjuvant taxane-based therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524
Dates: Start 1998-04; Study Completion 2003-10

PRIMARY OUTCOMES:
Time to disease progression with maintenance paclitaxel versus observation

SECONDARY OUTCOMES:
Overall survival
Toxicity
Quality of live
Conversion to a better response

CONTACTS AND LOCATIONS:
Overall Officials: PierFranco Conte, MD, Principal Investigator — University of Modena, Italy; Dino Amadori, MD, Principal Investigator — Morgagni-Pierantoni Hospital, Forli, Italy; Mario Delena, MD, Principal Investigator — Oncology Institute, Bari, Italy
Locations (7):
- Italy (7):
  - Azienda Ospedaliera Pisana, Pisa, PI
  - Oncology Institute, Bari
  - Morgagni-Pierantoni Hospital, Forlì
  - National Cancer Research Institute, Genoa
  - S. Carlo Hospital, Potenza
  - Santa Maria Nuova Hospital, Reggio Emilia
  - University of Rome, Rome